CLINICAL TRIAL: NCT04492670
Title: The Therapeutic Effect of a Combined Therapy of Tui-na and Oral Chinese Medicine on Osteoarthritis of Knee - A Randomized Wait-list Controlled Trial
Brief Title: Tui-na and Oral Chinese Medicine on KOA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Lin Zhixiu, Associate professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KOA
Record Dates: First submitted 2020-07-28; First posted 2020-07-30 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis, Tui-na, Chinese medicine
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tui-na and oral Chinese medicine (Experimental): 8 sessions of 20 minutes Tui-na for 4 weeks and take study medication (Herbal granules) twice daily concomitantly for 4weeks
  Interventions: Procedure: Tui-na; Drug: Du-Huo-Ji-Sheng-Tang (DHJST)
- Tui-na (Other): 8 sessions of 20 minutes Tui-na for 4 weeks
  Interventions: Procedure: Tui-na

INTERVENTIONS:
Procedure: Tui-na — For administering of Tui-na manipulation practice, responsible Tui-na CMP must have at least 2 years of clinical experience. The pre-trial workshops led by a senior practitioner will be organized to ensure standardization of Tui-na treatment manipulation and procedures.
Drug: Du-Huo-Ji-Sheng-Tang (DHJST) — This study medication is derived from Du-Huo-Ji-Sheng-Tang (DHJST) and concentrated Chinese Medicine granules will be used.
  Other Names: Herbal granules
  Arms: Tui-na and oral Chinese medicine

SUMMARY:
The study aims to evaluate the therapeutic effect of the Tui-na and oral Chinese medicine on the treatment of KOA.

This is a prospective, randomized wait-list controlled trial in patients with knee osteoarthritis (KOA). After 2 weeks screening period, eligible subjects will be randomly assigned to the treatment group and wait-list control group in 1:1 ratio. Subjects will have 4-week of treatment, and then a 4-week follow-up.

DETAILED DESCRIPTION:
The subjects will come for a screening visit at week 0 (baseline), then at week 2, week 4, and week 8 for Chinese medicine practitioner (CMP) investigators assessments. The Western Ontario and McMaster University Osteoarthritis index (WOMAC) and EQ-5D-5L will be assessed and filled up at different timepoints. The treatment group will receive both Tui-na and study medication and the wait-list control group will receive Tui-na alone. CMPs will provide consultation under Chinese medicine theory. Study medication compliance and adverse events will also be assessed at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. of either gender (female must have either sterilization done or menopause)
2. ≥50years of age
3. meet the criteria of KOA according to the American College of Rheumatology

   * Knee pain, and
   * Any 4 of the following,

     * ≥ 50 years of age
     * Less than 30 minutes of morning stiffness
     * Crepitus on active motion
     * Bony tenderness
     * Bony enlargement
     * No palpable warmth of synovium
     * Osteophytes (Radiographic findings)
4. with WOMAC score ≥ 39
5. with written informed consentform signed (for illiterate subjects, their next-of-kin or an impartial witness will sign with subjects' permission)

Exclusion Criteria:

1. Known knee pain caused by infection, malignant or autoimmune diseases
2. Knee surgery or arthroscopy in the past year
3. Chondroprotective or intra-articular injection in the past 4 months
4. Systemic corticoid treatment in the past 4 months
5. Taking anticoagulants, antiplatelets, corticosteroids, psychiatric drugs, hormones, antiarrhythmic drugs or diuretics drugs
6. Subject with uncontrolled hypertension
7. Local antiphlogistic treatment, acupuncture, physiotherapy in the past 2 weeks
8. Known history of mental disorder
9. Known history of serious acute organic disease
10. Renal or liver function impairment
11. Known allergy to or have drug interaction with the study herb

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-09-14 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
The Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 4 weeks
  to assess the condition of patients with KOA, the minimum score is 0 and maximum is 96

SECONDARY OUTCOMES:
EQ-5D-EL questionnaire | 8 weeks
  to assess health-related quality of life, one part is descriptive has 5 response level, the other part is VAS which ranges from 0 to 100
The Western Ontario and McMaster Universities Arthritis Index (WOMAC) | at 2 weeks and 8 weeks
  to assess the condition of patients with KOA, the minimum score is 0 and maximum is 96

CONTACTS AND LOCATIONS:
Overall Officials: Zhixiu Lin, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan KH, Ching JYL, Chan KL, Lau HY, Chu KM, Chan K, Pang HF, Wong LC, Chia CP, Zhang HW, Song T, Leung SB, Ng BFL, Lin ZX. Therapeutic effect of Duhuo Jisheng Decoction add-on Tui-na manipulation on osteoarthritis of knee: a randomized controlled trial. Chin Med. 2023 Jul 10;18(1):82. doi: 10.1186/s13020-023-00737-5. PMID 37424023